CLINICAL TRIAL: NCT07158008
Title: The SLEEVE-GERD Trial: A Comparative Study of Nissen-Sleeve and Roux-en-Y Gastric Bypass in Obese Patients With GERD
Brief Title: Comparison of Nissen-Sleeve and Gastric Bypass for GERD in Obese Patients
Acronym: SLEEVE-GERD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Michał Pędziwiatr, Chair of Surgery Department, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLEEVE-GERD Trial
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Gastro Esophageal Reflux; Severe Obesity; Bariatric Surgery
Keywords: Nissen-Sleeve; Gastric Bypass; GERD
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: Participants with obesity and gastroesophageal reflux disease (GERD) symptoms are randomly assigned in a 1:1 ratio to undergo either Nissen-Sleeve Gastrectomy (N-SG) or Roux-en-Y Gastric Bypass (RYGB). Randomization is stratified and block-based, with allocation concealed using sealed envelopes. A third, non-randomized observational cohort of patients without GERD undergoing standard sleeve gastrectomy (SG) is included to allow matched secondary analyses. The primary comparison is between the two randomized arms (N-SG vs. RYGB).
Masking Description: This is an open-label study. Due to the nature of the surgical interventions, masking of participants and healthcare providers is not feasible. Both the patients and the surgical team are aware of the assigned intervention. Outcome assessors and data analysts will be blinded during statistical analysis to minimize potential bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nissen-Sleeve Gastrectomy (N-SG) (Experimental): Participants in this arm will undergo laparoscopic sleeve gastrectomy combined with Nissen fundoplication. The procedure includes partial preservation of the gastric fundus to form a 360-degree wrap around the distal esophagus, followed by sleeve resection of the remaining stomach. This technique aims to provide both weight loss and reflux control while maintaining gastrointestinal continuity.
  Interventions: Procedure: Nissen-Sleeve Gastrectomy (N-SG)
- Roux-en-Y Gastric Bypass (RYGB) (Active Comparator): Participants in this arm will undergo standard laparoscopic Roux-en-Y gastric bypass. The procedure includes the creation of a small gastric pouch, a 100 cm alimentary (Roux) limb, and a 150 cm biliopancreatic limb. The bypass alters the gastrointestinal anatomy to promote weight loss and has established effectiveness in reducing GERD symptoms.
  Interventions: Procedure: Roux-en-Y Gastric Bypass (RYGB)
- Sleeve Gastrectomy - Control (No GERD) (Other): This non-randomized observational group includes patients without GERD symptoms undergoing standard sleeve gastrectomy. Data from this group will be used for secondary matched analyses to evaluate weight loss and hormonal changes, serving as a control for comparative evaluation with the randomized arms.
  Interventions: Procedure: Sleeve Gastrectomy (SG)

INTERVENTIONS:
Procedure: Nissen-Sleeve Gastrectomy (N-SG) — Laparoscopic Nissen-Sleeve Gastrectomy is a modification of standard sleeve gastrectomy that incorporates an anti-reflux procedure. The greater curvature of the stomach is mobilized and short gastric vessels are divided. A segment of the gastric fundus is preserved and passed behind the distal esophagus to create a 360-degree wrap (Nissen fundoplication) around the lower esophageal sphincter. The crura of the diaphragm are approximated if necessary. Following fundoplication, the remainder of the stomach is resected longitudinally over a 40 French bougie using a linear stapling device, creating a tubular gastric conduit. This approach aims to achieve weight loss while providing a functional anti-reflux barrier and maintaining gastrointestinal continuity.
  Arms: Nissen-Sleeve Gastrectomy (N-SG)
Procedure: Roux-en-Y Gastric Bypass (RYGB) — Laparoscopic Roux-en-Y Gastric Bypass is a standard bariatric procedure that combines gastric restriction with intestinal bypass. A small proximal gastric pouch is created using linear staplers, completely separating it from the gastric remnant. A 100 cm alimentary (Roux) limb of jejunum is measured from the ligament of Treitz and anastomosed to the gastric pouch (gastrojejunostomy) using a linear stapler. A jejunojejunostomy is then performed 150 cm distal to the gastrojejunostomy to connect the biliopancreatic limb to the alimentary limb, restoring intestinal continuity. The mesenteric defects are closed to reduce the risk of internal hernia. This procedure promotes weight loss and has established effectiveness in reducing gastroesophageal reflux symptoms.
  Arms: Roux-en-Y Gastric Bypass (RYGB)
Procedure: Sleeve Gastrectomy (SG) — Laparoscopic Sleeve Gastrectomy is a restrictive bariatric procedure involving longitudinal resection of the stomach to create a tubular gastric conduit. The greater curvature is mobilized and short gastric vessels are divided. Using a bougie as a guide, the stomach is divided with a linear stapling device from the antrum to the angle of His, removing approximately 75-80% of gastric volume, including most of the fundus. This reduces stomach capacity and ghrelin production, promoting weight loss while maintaining gastrointestinal continuity.
  Arms: Sleeve Gastrectomy - Control (No GERD)

SUMMARY:
This randomized clinical trial aims to compare two surgical techniques for the treatment of obesity in patients who also have symptoms of gastroesophageal reflux disease (GERD). The study will compare Nissen-Sleeve Gastrectomy (N-SG)-a sleeve gastrectomy combined with a reflux-preventing procedure-to the Roux-en-Y Gastric Bypass (RYGB), which is the current standard surgical option for obese patients with GERD.

Both procedures are widely used to treat severe obesity, but they differ in how they affect the digestive system and the potential for reflux control, nutritional outcomes, and future surgical options. N-SG is a newer technique that preserves the natural pathway of the gastrointestinal tract and allows standard endoscopic access to the bile ducts, which may be beneficial for long-term patient care. RYGB, on the other hand, bypasses part of the stomach and small intestine, which may lead to better reflux resolution but carries risks of nutritional deficiencies and altered anatomy.

Eligible participants with obesity and GERD symptoms will be randomly assigned to receive either N-SG or RYGB. The primary goal is to evaluate whether N-SG is not inferior to RYGB in reducing GERD symptoms one year after surgery. Secondary outcomes include weight loss, quality of life, surgical complications, and changes in the hormone ghrelin, which is involved in appetite regulation.

In addition, a larger control group of patients without GERD undergoing standard sleeve gastrectomy will be recruited to allow further comparisons. All participants will be followed for one year after surgery, with blood samples, questionnaires, and clinical data collected to assess both metabolic and reflux-related outcomes.

This study is being conducted at the University Hospital in Kraków, Poland, and aims to improve the personalization of bariatric treatment for patients suffering from both obesity and reflux.

DETAILED DESCRIPTION:
This randomized clinical trial is designed to compare the safety and effectiveness of Nissen-Sleeve Gastrectomy (N-SG) versus Roux-en-Y Gastric Bypass (RYGB) in patients with obesity and symptoms of gastroesophageal reflux disease (GERD). N-SG is a modified sleeve gastrectomy procedure that incorporates an anti-reflux mechanism based on the Nissen fundoplication technique, while RYGB is a well-established bariatric procedure with proven anti-reflux efficacy.

Background and Rationale:

Severe obesity (BMI ≥ 40 or ≥ 35 with comorbidities) is a growing health problem and is frequently associated with GERD. While sleeve gastrectomy (SG) is currently the most widely performed bariatric procedure globally, it has been associated with the development or worsening of GERD in a significant number of cases. RYGB has become the standard surgical approach in obese patients with pre-existing GERD due to its high rate of reflux symptom resolution. However, RYGB involves more complex anatomical changes, carries a risk of nutritional deficiencies, and limits future endoscopic access to the biliary tract.

The Nissen-Sleeve Gastrectomy (N-SG), first described by David Nocca in 2016, combines SG with a 360-degree gastric fundoplication wrap (similar to that used in traditional Nissen fundoplication). This technique preserves gastrointestinal continuity and potentially maintains endoscopic access to the duodenum, while adding a reflux barrier. Early observational studies suggest favorable outcomes in terms of GERD resolution while retaining the benefits of SG. However, no large-scale randomized controlled trial has compared N-SG with RYGB in this specific patient population.

Study Design:

This is a prospective, single-center, randomized controlled non-inferiority trial conducted at the University Hospital in Kraków, Poland. Patients with obesity and clinically confirmed GERD will be randomized in a 1:1 ratio to receive either N-SG or RYGB. Randomization is performed using a computer-generated block randomization schedule. Allocation will be concealed in sealed envelopes and opened immediately prior to surgery. The estimated sample size for the randomized arms is 140 patients (70 per group), accounting for an assumed 15% dropout rate, and powered to detect non-inferiority with a margin of 10%.

In addition to the randomized comparison, a non-randomized observational control group of approximately 420 patients undergoing standard SG without GERD symptoms will be enrolled. This group will allow propensity-matched analyses and further comparisons of outcomes.

Surgical Techniques:

Nissen-Sleeve Gastrectomy (N-SG): The greater curvature of the stomach is mobilized, short gastric vessels are divided, and the fundus is used to create a posterior wrap around the distal esophagus. A 360-degree fundoplication (Nissen) is performed laparoscopically. This is followed by longitudinal gastric resection using a 40Fr bougie to calibrate the sleeve.

Roux-en-Y Gastric Bypass (RYGB): A small proximal gastric pouch is created. A 100 cm alimentary (Roux) limb is anastomosed to the pouch. A biliopancreatic limb of 150 cm is created via jejunojejunostomy, and the continuity of the gastrointestinal tract is restored. The stomach remnant and duodenum are excluded from the alimentary flow.

Follow-Up and Data Collection:

All patients will be followed for at least 12 months postoperatively. Clinical data will be collected at baseline, postoperatively, and at follow-up visits. Blood samples will be obtained at four time points: (1) day of surgery, (2) first postoperative day, (3) one week post-discharge (during suture removal), and (4) at 12-month follow-up. Blood will be analyzed for serum ghrelin levels using ELISA-based testing.

GERD symptoms will be assessed pre- and postoperatively using the validated GerdQ questionnaire. A score below 5 at 12 months, along with discontinuation of proton pump inhibitor (PPI) therapy for at least 60 days, will be considered remission of GERD.

Outcomes:

Primary outcome: GERD symptom resolution at 12 months post-op, comparing N-SG to RYGB.

Secondary outcomes: Weight loss (measured as %EWL, %TWL, and BMI change), serum ghrelin levels, incidence of postoperative complications (Clavien-Dindo scale), and quality of life metrics.

Control Group:

Patients without GERD undergoing standard SG will serve as an observational control cohort. This group will provide comparative data on weight loss and metabolic changes without the influence of pre-existing reflux disease. Their data will be used for secondary analyses and matched comparisons.

Ethical Considerations:

The study has received approval from the Bioethics Committee of Jagiellonian University Medical College. Written informed consent will be obtained from all participants. Participation is voluntary, and subjects may withdraw at any time. The N-SG technique is investigational in Poland and may only be offered within this trial framework. Patients declining randomization will receive the standard of care (RYGB or SG based on clinical indication).

Potential Risks and Complications:

Both RYGB and SG are well-established surgical procedures. N-SG may be associated with additional risks specific to fundoplication, such as cuff leak or stenosis. These complications will be managed with standard endoscopic or surgical protocols as needed. All participants will be closely monitored throughout the study.

This trial seeks to evaluate whether N-SG can offer equivalent reflux control to RYGB while avoiding the anatomical disruption and long-term risks associated with bypass surgery. The results may support broader adoption of N-SG as a tailored option for obese patients with GERD.

ELIGIBILITY:
Inclusion Criteria:

For N-Sleeve Gastrectomy (N-SG) and Roux-en-Y Gastric Bypass (RYGB) arms:

* Age ≥ 18 years
* Written informed consent provided
* Eligible for bariatric surgery according to national guidelines (BMI ≥ 40 kg/m² or BMI ≥ 35 kg/m² with obesity-related comorbidities)
* Presence of symptomatic gastroesophageal reflux disease (GERD), defined by at least one of the following:
* Regular use of proton pump inhibitors (PPIs)
* GerdQ score > 6
* Endoscopic evidence of esophagitis (Los Angeles classification grade B or higher)

For Sleeve Gastrectomy (SG) observational control group:

* Age ≥ 18 years
* Written informed consent provided
* Eligible for bariatric surgery according to national guidelines (BMI ≥ 40 kg/m² or BMI ≥ 35 kg/m² with obesity-related comorbidities)
* No symptoms or history of GERD

Exclusion Criteria:

* History of prior anti-reflux surgery
* History of upper gastrointestinal tract surgery
* Active smoking or history of nicotine use
* Severe cardiac insufficiency (New York Heart Association Class III or IV)
* Pregnancy or planned pregnancy during the study period (if applicable based on future additions)
* Any condition that, in the opinion of the investigator, would interfere with the participant's ability to comply with the study protocol or would pose additional risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
GERD Symptom Remission | 12 months post-surgery
  Resolution of GERD symptoms, defined as:
  No need for proton pump inhibitors (PPIs) for at least 60 consecutive days, and
  GerdQ questionnaire score < 7 at 12-month follow-up. Comparison between Nissen-Sleeve Gastrectomy (N-SG) and Roux-en-Y Gastric Bypass (RYGB) arms.

SECONDARY OUTCOMES:
Percent Excess Weight Loss (%EWL) | 12 months post-surgery
  Percentage of excess weight loss, calculated based on initial excess body weight. Compared across all three study arms.
Percent Total Weight Loss (%TWL) | 12 months post-surgery
  Percentage of total body weight loss from baseline. Compared across all three study arms.
Change in Body Mass Index (BMI) | Difference in BMI from baseline to 12 months. Compared across all three study arms.
  12 months post-surgery
Change in Serum Ghrelin Levels | Baseline (day of surgery), postoperative day 1, day 7 after discharge, and 12 months post-surgery
  Change in fasting plasma ghrelin concentration measured by ELISA assay. Compared across N-SG, RYGB, and SG (control) arms.
Postoperative Complication Rate (Clavien-Dindo Classification ≥ Grade III) | Up to 30 days post-surgery
  Number and percentage of serious postoperative complications classified as Clavien-Dindo grade III or higher.
Quality of Life (QoL) Score | 12 months post-surgery
  Quality of life assessed using validated tools (BAROS) Comparison between N-SG and RYGB arms.
GERD Related Quality of Life | 12 months post-surgery
  Assesment of changes in quality of life associated with GERD using GERD-HRQL questionnaire comparing N-SG with RYGB before surgery and 12 months after

CONTACTS AND LOCATIONS:
Locations (1):
- Szpital Uniwersytecki w Krakowie, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Yes
IPD to Be Shared: De-identified individual-level data related to primary and secondary outcomes, including weight loss metrics, GERD scores, and hormone levels.
  When Available: 12 months after publication of primary results How Long Available: For 3 years after results publication With Whom: Qualified researchers upon request Access Criteria: Requests must include a methodologically sound proposal and data use agreement. Data will be shared via institutional data-sharing platform or secure transfer.
  For What Types of Analyses: For academic, non-commercial research related to obesity, bariatric surgery, and GERD outcomes